CLINICAL TRIAL: NCT01328158
Title: Drug Use Investigation of Kaletra Tablets (Quaque Die, QD) on Patients With HIV-infection
Brief Title: Drug Use Investigation of Kaletra Tablets (Once Daily Administration) on Patients With HIV-infection
Status: Completed | Type: Observational
Sponsor: AbbVie (prior sponsor, Abbott) (Industry)
Responsible Party: Sponsor
Organization: AbbVie (Industry)
Other Study IDs: P12-760
Record Dates: First submitted 2011-04-01; First posted 2011-04-04 (Estimated); Results first posted 2014-12-22 (Estimated); Last update posted 2014-12-22 (Estimated); Status verified 2014-12

CONDITIONS: Human Immunodeficiency Virus Infection
Keywords: Kaletra, Lopinavir (LPV)/Ritonavir (RTV), Human Immunodeficiency Virus (HIV) infection
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Lopinavir/Ritonavir: Participants with HIV infection who were receiving Lopinavir/Ritonavir or who started Lopinavir/Ritonavir therapy during the registration period were evaluated

SUMMARY:
This study of Kaletra (Lopinavir (LPV)/Ritonavir (RTV)) tablets will be conducted to clarify the following with regard to treatment with this drug:

1. Incidence and conditions of occurrence of adverse reactions in the clinical setting
2. Factors that may affect the safety and effectiveness of Kaletra (QD)

ELIGIBILITY:
Inclusion Criteria:

- Participants who were receiving Kaletra or who started Kaletra therapy during the registration period.

Exclusion Criteria:

* Participants with a history of hypersensitivity to any ingredient of this drug.
* Participants who are undergoing treatment with any of the following drugs: pimozide, ergotamine tartrate, dihydroergotamine mesilate, ergometrine maleate, methylergometrine maleate, midazolam, triazolam, vardenafil hydrochloride hydrate, sildenafil citrate (Revatio), tadalafil (Adcirca), blonanserin, azelnidipine, rivaroxaban, voriconazole.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All participants who receive Kaletra for the treatment of Human Immunodeficiency Virus infection per approved label
Sampling Method: Non-Probability Sample
Enrollment: 236 (Actual)
Dates: Start 2011-06; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susumu Adachi, MD, Study Director — AbbVie G.K.
Locations (23):
- Japan (23):
  - Site Reference ID/Investigator# 57629, Fukuoka
  - Site Reference ID/Investigator# 57630, Hiroshima
  - Site Reference ID/Investigator# 57631, Hokkaido
  - Site Reference ID/Investigator# 57628, Kitakyushu-shi
  - Site Reference ID/Investigator# 57638, Kurashiki-shi
  - Site Reference ID/Investigator# 57634, Kyoto
  - Site Reference ID/Investigator# 57625, Nagoya
  - Site Reference ID/Investigator# 57626, Nagoya
  - Site Reference ID/Investigator# 57637, Niigata
  - Site Reference ID/Investigator# 57632, Nishinomiya-shi
  - Site Reference ID/Investigator# 57639, Osaka
  - Site Reference ID/Investigator# 57640, Osaka
  - Site Reference ID/Investigator# 57636, Sendai
  - Site Reference ID/Investigator# 48722, Tokyo
  - Site Reference ID/Investigator# 57641, Tokyo
  - Site Reference ID/Investigator# 57643, Tokyo
  - Site Reference ID/Investigator# 57644, Tokyo
  - Site Reference ID/Investigator# 57645, Tokyo
  - Site Reference ID/Investigator# 57646, Tokyo
  - Site Reference ID/Investigator# 57647, Tokyo
  - Site Reference ID/Investigator# 57648, Tokyo
  - Site Reference ID/Investigator# 57650, Tokyo
  - Site Reference ID/Investigator# 57633, Yokohama

REFERENCES:
- See also: Related Info — http://rxabbvie.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Survey forms were collected from 236 patients. 16 participants completed treatment with Lopinavir/Ritonavir tablets before the start of enrollment in this study and were excluded from the analysis.
Period: Overall Study
Arm/Group | Lopinavir/Ritonavir
Started | 220
Completed | 220
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: All participants who received Lopinavir/Ritonavir for the treatment of HIV infection in institutions participating in the HRD Cooperative Survey during the registration period.
Arm/Group | Lopinavir/Ritonavir
Number analyzed (Participants) | 220
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.6 (10.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 205
Presence/Absence of Previous Treatment of HIV-Infection [Number; unit: participants]
  Absent | 10
  Present | 210

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Adverse Drug Reactions
Description: Adverse Drug Reactions are adverse events for which relationship with Lopinavir/Ritonavir tablets is considered as "Related", "Relationship cannot be ruled out", and "Unknown".
Time Frame: Up to 60 Months
Population: as for baseline characteristics
Measure: Number; unit: percentage of participants
Arm/Group | Lopinavir/Ritonavir
Number analyzed (Participants) | 220
percentage of participants | 37.73

2. Primary Outcome: Number of Adverse Drug Reactions
Description: as for outcome 1
Time Frame: Up to 60 Months
Population: as for baseline characteristics
Measure: Number; unit: number of adverse drug reaction
Arm/Group | Lopinavir/Ritonavir
Number analyzed (Participants) | 220
number of adverse drug reaction | 124

3. Secondary Outcome: Number of Participants With Adverse Drug Reaction by Patient Characteristic: Gender
Description: Participants with adverse drug reactions were assessed in this study. Adverse Drug Reactions are adverse events for which relationship with Lopinavir/Ritonavir tablets is considered as "Related", "Relationship cannot be ruled out", and "Unknown".
Time Frame: Up to 60 Months
Population: as for baseline characteristics
Measure: Number; unit: participants
Arm/Group | Lopinavir/Ritonavir
Number analyzed (Participants) | 220
participants
  Male (n=205) | 79
  Female (n=15) | 4

4. Secondary Outcome: Number of Participants With Adverse Drug Reaction by Patient Characteristic: Presence/Absence of Pregnancy
Description: as for outcome 3
Time Frame: Up to 60 Months
Population: All female participants who received Lopinavir/Ritonavir for the treatment of HIV infection in institutions participating in the HRD Cooperative Survey during the registration period.
Measure: Number; unit: participants
Arm/Group | Lopinavir/Ritonavir
Number analyzed (Participants) | 15
participants
  Absence of pregnancy (n=10) | 3
  Presence of pregnancy (n=5) | 1

5. Secondary Outcome: Number of Participants With Adverse Drug Reaction by Patient Characteristic: Age
Description: as for outcome 3
Time Frame: Up to 60 Months
Population: as for baseline characteristics
Measure: Number; unit: participants
Arm/Group | Lopinavir/Ritonavir
Number analyzed (Participants) | 220
participants
  ≤ 14 Years (n=0) | 0
  15 Years to ≤ 29 Years (n=10) | 3
  30 Years to ≤ 49 Years (n=158) | 62
  50 years to ≤ 64 Years (n=43) | 15
  ≥ 65 Years (n=8) | 3
  Unknown/Undescribed (n=1) | 0

6. Secondary Outcome: Number of Participants With Adverse Drug Reaction by Patient Characteristic: Inpatient/Outpatient
Description: as for outcome 3
Time Frame: Up to 60 Months
Population: as for baseline characteristics
Measure: Number; unit: participants
Arm/Group | Lopinavir/Ritonavir
Number analyzed (Participants) | 220
participants
  Inpatient (n=2) | 1
  Outpatient (n=191) | 74
  Switching between Inpatient and Outpatient (n=27) | 8

7. Secondary Outcome: Number of Participants With Adverse Drug Reaction by Patient Characteristic: Presence/Absence of Previous Treatment of Human Immunodeficiency Virus (HIV)-Infection
Description: as for outcome 3
Time Frame: Up to 60 Months
Population: as for baseline characteristics
Measure: Number; unit: participants
Arm/Group | Lopinavir/Ritonavir
Number analyzed (Participants) | 220
participants
  Absent (n=10) | 1
  Present (n=210) | 82

8. Secondary Outcome: Number of Participants With Adverse Drug Reaction by Patient Characteristic: Races
Description: as for outcome 3
Time Frame: Up to 60 Months
Population: as for baseline characteristics
Measure: Number; unit: participants
Arm/Group | Lopinavir/Ritonavir
Number analyzed (Participants) | 220
participants
  Japanese (n=204) | 74
  Other (n=16) | 9

9. Secondary Outcome: Number of Participants With Adverse Drug Reaction by Patient Characteristic: Route of Infection
Description: as for outcome 3
Time Frame: Up to 60 Months
Population: as for baseline characteristics
Measure: Number; unit: participants
Arm/Group | Lopinavir/Ritonavir
Number analyzed (Participants) | 220
participants
  Blood Product (n=17) | 5
  Mother-to-Child Transmission (n=0) | 0
  Medical Accident (n=0) | 0
  Other (n=179) | 70
  Unknown/Undescribed (n=24) | 8

10. Secondary Outcome: Number of Participants With Adverse Drug Reaction by Patient Characteristic: Disease Duration
Description: as for outcome 3
Time Frame: Up to 60 Months
Population: as for baseline characteristics
Measure: Number; unit: participants
Arm/Group | Lopinavir/Ritonavir
Number analyzed (Participants) | 220
participants
  ≤ 1 Year (n=0) | 0
  1 Year to ≤ 2 Years (n=0) | 0
  2 Years to ≤ 3 Years (n=2) | 0
  3 Years to ≤ 4 Years (n=1) | 0
  4 Years to ≤ 5 Years (n=2) | 1
  >5 Years (n=10) | 6
  Unknown/Undescribed (n=205) | 76

11. Secondary Outcome: Number of Participants With Adverse Drug Reaction by Patient Characteristic: Presence/Absence of Past Medical History
Description: as for outcome 3
Time Frame: Up to 60 Months
Measure: Number; unit: participants
Arm/Group | Lopinavir/Ritonavir
Number analyzed (Participants) | 220
participants
  Absent (n=77) | 24
  Present (n=137) | 56
  Unknown/Undescribed (n=6) | 3

12. Secondary Outcome: Number of Participants With Adverse Drug Reaction by Patient Characteristic: Presence/Absence of Allergy
Description: as for outcome 3
Time Frame: Up to 60 Months
Population: as for baseline characteristics
Measure: Number; unit: participants
Arm/Group | Lopinavir/Ritonavir
Number analyzed (Participants) | 220
participants
  Absent (n=135) | 41
  Present (n=67) | 35
  Unknown/Undescribed (n=18) | 7

13. Secondary Outcome: Number of Participants With Adverse Drug Reaction by Patient Characteristic: Presence/Absence of Concomitant Diseases
Description: as for outcome 3
Time Frame: Up to 60 Months
Population: as for baseline characteristics
Measure: Number; unit: participants
Arm/Group | Lopinavir/Ritonavir
Number analyzed (Participants) | 220
participants
  Absent (n=52) | 14
  Present (n=168) | 69

14. Secondary Outcome: Number of Participants With Adverse Drug Reaction by Patient Characteristic: Presence/Absence of Concomitant Renal Disorder
Description: as for outcome 3
Time Frame: Up to 60 Months
Population: as for baseline characteristics
Measure: Number; unit: participants
Arm/Group | Lopinavir/Ritonavir
Number analyzed (Participants) | 220
participants
  Absent (n=217) | 82
  Present (n=3) | 1

15. Secondary Outcome: Number of Participants With Adverse Drug Reaction by Patient Characteristic: Presence/Absence of Concomitant Liver Disorder
Description: as for outcome 3
Time Frame: Up to 60 Months
Population: as for baseline characteristics
Measure: Number; unit: participants
Arm/Group | Lopinavir/Ritonavir
Number analyzed (Participants) | 220
participants
  Absent (n=159) | 60
  Present (n=61) | 23
  Hepatitis Present (n=49) | 18

16. Secondary Outcome: Number of Participants With Adverse Drug Reaction by Patient Characteristic: Haemophilia
Description: as for outcome 3
Time Frame: Up to 60 Months
Population: as for baseline characteristics
Measure: Number; unit: participants
Arm/Group | Lopinavir/Ritonavir
Number analyzed (Participants) | 220
participants
  Absent (n=203) | 78
  Haemophilia A: Present (n=11) | 4
  Haemophilia B: Present (n=6) | 1

17. Secondary Outcome: Number of Participants With Adverse Drug Reaction by Patient Characteristic: Haemophilia With/Without Hepatitis C
Description: as for outcome 3
Time Frame: Up to 60 Months
Population: as for baseline characteristics
Measure: Number; unit: participants
Arm/Group | Lopinavir/Ritonavir
Number analyzed (Participants) | 17
participants
  Without Hepatitis C (n=3) | 0
  With Hepatitis C (n=14) | 5

18. Secondary Outcome: Number of Participants With Adverse Drug Reaction by Patient Characteristic: Center for Disease Control (CDC) Classification Category of Severity Before Treatment
Description: as for outcome 3
Time Frame: Up to 60 Months
Population: as for baseline characteristics
Measure: Number; unit: participants
Arm/Group | Lopinavir/Ritonavir
Number analyzed (Participants) | 220
participants
  A (n=9) | 2
  B (n=0) | 0
  C (n=5) | 0
  P-0 (n=0) | 0
  P-1 (n=0) | 0
  P-2 (n=0) | 0
  Unknown/Undescribed (n=206 | 81

19. Secondary Outcome: Number of Participants With Adverse Drug Reaction by Patient Characteristic: Administration Method of Lopinavir/Ritonavir
Description: as for outcome 3
Time Frame: Up to 60 Months
Population: as for baseline characteristics
Measure: Number; unit: participants
Arm/Group | Lopinavir/Ritonavir
Number analyzed (Participants) | 220
participants
  2 Tabs × 2 Times/Day (n=156) | 63
  4 Tabs × 1 Time/Day (n=56) | 17
  2 × 2 Changing to 4 x 1 Tabs x Times/Day (n=5) | 1
  Switch Between 2x2 and 4x1 Tabs x Times/Day (n=0) | 0
  Other (3 Tabs x 2 Times as Other Daily Dose) (n=2) | 2
  Unknown/Undescribed (n=1) | 0

20. Secondary Outcome: Number of Participants With Adverse Drug Reaction by Patient Characteristic: Mean Daily Dose of Lopinavir/Ritonavir
Description: as for outcome 3
Time Frame: Up to 60 Months
Population: as for baseline characteristics
Measure: Number; unit: participants
Arm/Group | Lopinavir/Ritonavir
Number analyzed (Participants) | 220
participants
  < Lopinavir 800/Ritonavir 200 mg (n=0) | 0
  Lopinavir 800/Ritonavir 200 mg (n=217) | 81
  > Lopinavir 800/Ritonavir 200 mg (n=3) | 2

21. Secondary Outcome: Number of Participants With Adverse Drug Reaction by Patient Characteristic: Use Duration of Lopinavir/Ritonavir
Description: as for outcome 3
Time Frame: Up to 60 Months
Population: as for baseline characteristics
Measure: Number; unit: participants
Arm/Group | Lopinavir/Ritonavir
Number analyzed (Participants) | 220
participants
  ≤ 30 Days (n=5) | 1
  31 Days to ≤ 180 Days (n=27) | 13
  181 Days to ≤ 364 Days (n=19) | 9
  ≥ 365 Days (n=168) | 60
  Unknown/Undescribed (n=1) | 0

22. Secondary Outcome: Number of Participants With Adverse Drug Reaction by Patient Characteristic: Presence/Absence of Anti-HIV Concomitant Drugs
Description: as for outcome 3
Time Frame: Up to 60 Months
Population: as for baseline characteristics
Measure: Number; unit: participants
Arm/Group | Lopinavir/Ritonavir
Number analyzed (Participants) | 220
participants
  Absent (n=0) | 0
  Present (n=220) | 83

23. Secondary Outcome: Number of Participants With Adverse Drug Reaction by Patient Characteristic: Presence/Absence of Anti-HIV Concomitant Non-Drug Treatments
Description: as for outcome 3
Time Frame: Up to 60 Months
Population: as for baseline characteristics
Measure: Number; unit: participants
Arm/Group | Lopinavir/Ritonavir
Number analyzed (Participants) | 220
participants
  Absent (n=206) | 76
  Present (n=14) | 7

24. Secondary Outcome: Number of Participants With Adverse Drug Reaction by Patient Characteristic: Types of Concomitant Anti-HIV Drugs
Description: Participants with adverse drug reactions were assessed in this study. Adverse Drug Reactions are adverse events for which relationship with Lopinavir/Ritonavir tablets is considered as "Related", "Relationship cannot be ruled out", and "Unknown". Abbreviations for the following terminologies are used to represent results in below table: NRTIs: Nucleoside Reverse Transcriptase Inhibitors, NNRTIs: Non-Nucleoside Reverse Transcriptase Inhibitors.
Time Frame: Up to 60 Months
Population: as for baseline characteristics
Measure: Number; unit: participants
Arm/Group | Lopinavir/Ritonavir
Number analyzed (Participants) | 220
participants
  NRTIs (n=214 | 81
  NNRTIs (n=9) | 6
  Integrase Inhibitors (n=11) | 3
  CCR5 Inhibitors (n=0) | 0

25. Secondary Outcome: Number of Participants With Adverse Drug Reaction by Patient Characteristic: Presence/Absence of Concomitant Drugs Other Than Anti-HIV Drugs
Description: as for outcome 3
Time Frame: Up to 60 Months
Population: as for baseline characteristics
Measure: Number; unit: participants
Arm/Group | Lopinavir/Ritonavir
Number analyzed (Participants) | 220
participants
  Absent (n=104) | 29
  Present (n=116) | 54

26. Secondary Outcome: Number of Participants With Serious Adverse Events
Description: A serious adverse event is an adverse event that 1. requires in patient hospitalization or prolongation of existing hospitalization, 2. results in persistent or significant disability/incapacity, 3. is life-threatening, 4. results in death, 5. is a congenital anomaly/birth defect, or 6. is an important medical event other than the above.
Time Frame: Up to 60 Months
Population: as for baseline characteristics
Measure: Number; unit: participants
Arm/Group | Lopinavir/Ritonavir
Number analyzed (Participants) | 220
participants | 20

27. Secondary Outcome: Mean Cluster of Differentiation 4 (CD4) Cell Count in Treatment-Naive Participants at Each Time Point of Observation
Time Frame: Months 0, 3, 6, 9, 12, 24, 36, 48, and 60 after first dosing of Lopinavir/Ritonavir
Population: Participants who had both a baseline and at least one post-baseline CD4 cell count value were included in the effectiveness analysis set.
Measure: Mean (Standard Deviation); unit: cells/mm^3
Arm/Group | Lopinavir/Ritonavir
Number analyzed (Participants) | 6
cells/mm^3
  Use Duration: 0 Months (n=6) | 144.5 (130.9)
  Use Duration: 3 Months (n=0) | NA (NA) — No data available for assessment.
  Use Duration: 6 Months (n=1) | 190.0 (NA) — Standard Deviation cannot be calculated as CD4 cell count is available for 1 subject only.
  Use Duration: 9 Months (n=0) | NA (NA) — No data available for assessment.
  Use Duration: 12 Months (n=1) | 104.0 (NA) — Standard Deviation cannot be calculated as CD4 cell count is available for 1 subject only.
  Use Duration: 24 Months (n=3) | 184.3 (225.4)
  Use Duration: 36 Months (n=2) | 330.0 (200.8)
  Use Duration: 48 Months (n=1) | 474.0 (NA) — Standard Deviation cannot be calculated as CD4 cell count is available for 1 subject only.
  Use Duration: 60 Months (n=1) | 377.0 (NA) — Standard Deviation cannot be calculated as CD4 cell count is available for 1 subject only.

28. Secondary Outcome: Mean CD4 Cell Count in Treatment-Experienced Participants at Each Time Point of Observation
Time Frame: Months 0, 3, 6, 9, 12, 24, 36, 48, and 60 after first dosing of Lopinavir/Ritonavir
Population: as for outcome 27
Measure: Mean (Standard Deviation); unit: cells/mm^3
Arm/Group | Lopinavir/Ritonavir
Number analyzed (Participants) | 4
cells/mm^3
  Use Duration: 0 Months (n=4) | 654.5 (280.4)
  Use Duration: 3 Months (n=1) | 657.0 (NA) — Standard Deviation cannot be calculated as CD4 cell count is available for 1 subject only.
  Use Duration: 6 Months (n=1) | 835.0 (NA) — Standard Deviation cannot be calculated as CD4 cell count is available for 1 subject only.
  Use Duration: 9 Months (n=2) | 713.5 (82.7)
  Use Duration: 12 Months (n=2) | 878.5 (229.8)
  Use Duration: 24 Months (n=0) | NA (NA) — No data available for assessment.
  Use Duration: 36 Months (n=0) | NA (NA) — No data available for assessment.
  Use Duration: 48 Months (n=0) | NA (NA) — No data available for assessment.
  Use Duration: 60 Months (n=0) | NA (NA) — No data available for assessment.

29. Secondary Outcome: Mean HIV Ribonucleic Acid (RNA) Amount in Treatment-Naive Participants at Each Time Point of Observation
Description: For subjects with plasma HIV-1 RNA quantified as < 400 copies/mL, the result was recorded as 399 copies/mL.
Time Frame: Months 0, 3, 6, 9, 12, 24, 36, 48, and 60 after first dosing of Lopinavir/Ritonavir
Population: Participants who had both a baseline and at least one post-baseline HIV RNA value were included in the effectiveness analysis set.
Measure: Mean (Standard Deviation); unit: Log10 copies/mL
Arm/Group | Lopinavir/Ritonavir
Number analyzed (Participants) | 6
Log10 copies/mL
  Use Duration: 0 Months (n=6) | 5.2 (0.8)
  Use Duration: 3 Months (n=0) | NA (NA) — No data available for assessment.
  Use Duration: 6 Months (n=1) | 2.6 (NA) — Standard Deviation cannot be calculated as HIV-RNA value is available for 1 subject only.
  Use Duration: 9 Months (n=0) | NA (NA) — No data available for assessment.
  Use Duration: 12 Months (n=1) | 2.6 (NA) — Standard Deviation cannot be calculated as HIV-RNA value is available for 1 subject only.
  Use Duration: 24 Months (n=3) | 3.4 (1.3)
  Use Duration: 36 Months (n=2) | 2.6 (NA) — Standard Deviation cannot be calculated as HIV-RNA value is available for 1 subject only.
  Use Duration: 48 Months (n=1) | 2.6 (NA) — Standard Deviation cannot be calculated as HIV-RNA value is available for 1 subject only.
  Use Duration: 60 Months (n=1) | 2.6 (NA) — Standard Deviation cannot be calculated as HIV-RNA value is available for 1 subject only.

30. Secondary Outcome: Mean HIV RNA Amount in Treatment-Experienced Participants at Each Time Point of Observation
Description: For subjects with plasma HIV-1 RNA quantified as < 400 copies/mL, the result was recorded as 399 copies/mL.
Time Frame: Months 0, 3, 6, 9, 12, 24, 36, 48, and 60 after first dosing of Lopinavir/Ritonavir
Population: as for outcome 29
Measure: Mean (Standard Deviation); unit: Log10 copies/mL
Arm/Group | Lopinavir/Ritonavir
Number analyzed (Participants) | 4
Log10 copies/mL
  Use Duration: 0 Months (n=4) | 2.6 (0.0)
  Use Duration: 3 Months (n=1) | 2.6 (NA) — Standard Deviation cannot be calculated as HIV-RNA value is available for 1 subject only.
  Use Duration: 6 Months (n=1) | 2.6 (NA) — Standard Deviation cannot be calculated as HIV-RNA value is available for 1 subject only.
  Use Duration: 9 Months (n=2) | 2.6 (0.0)
  Use Duration: 12 Months (n=2) | 2.6 (0.0)
  Use Duration: 24 Months (n=0) | NA (NA) — No data available for assessment.
  Use Duration: 36 Months (n=0) | NA (NA) — No data available for assessment.
  Use Duration: 48 Months (n=0) | NA (NA) — No data available for assessment.
  Use Duration: 60 Months (n=0) | NA (NA) — No data available for assessment.

31. Secondary Outcome: Number of Participants in Each CDC Classification Category of HIV-infection Over Time
Description: CDC Categories include Category A: asymptomatic acute phase, Category B: symptomatic other than A or C, and Category C: having an AIDS-indicator disease.
Time Frame: Up to Month 60 after first dose of Lopinavir/Ritonavir
Population: as for baseline characteristics
Measure: Number; unit: participants
Groups:
- Lopinavir/Ritonavir: Baseline CDC Category A; Lopinavir/Ritonavir: Baseline CDC Category C; Lopinavir/Ritonavir: Baseline CDC Category Unknown: Participants with HIV infection who were receiving Lopinavir/Ritonavir or who started Lopinavir/Ritonavir therapy during the registration period were evaluated
Arm/Group | Lopinavir/Ritonavir: Baseline CDC Category A | Lopinavir/Ritonavir: Baseline CDC Category C | Lopinavir/Ritonavir: Baseline CDC Category Unknown
Number analyzed (Participants) | 9 | 5 | 206
participants
  CDC Category A After Treatment | 4 | 0 | 39
  CDC Category B After Treatment | 0 | 0 | 9
  CDC Category C After Treatment | 0 | 3 | 36
  CDC Category Unknown After Treatment | 5 | 2 | 122

32. Secondary Outcome: Percentage of Participants With Plasma HIV-1 RNA Levels Less Than 400 Copies/Milliliter [mL]) by Duration in Treatment-Naive Participants
Description: Participants whose number of plasma HIV-1 RNA copies was less than 400 copies/mL after the start of treatment were handled as responders. For subjects with plasma HIV-1 RNA quantified as < 400 copies/mL, the result was recorded as 399 copies/mL.
Time Frame: Months 0, 3, 6, 9, 12, 24, 36, 48, and 60 after first dosing of Lopinavir/Ritonavir
Population: Participants who had both a baseline and at least one post-baseline HIV-1 RNA value were included in the effectiveness analysis set.
Measure: Number; unit: percentage of participants
Arm/Group | Lopinavir/Ritonavir
Number analyzed (Participants) | 6
percentage of participants
  At 0 Months (n=6) | 0.0
  At 3 Months (n=0) | NA — No data available for assessment.
  At 6 Months (n=1) | 100.0
  AT 9 Months (n=0) | NA — No data available for assessment.
  At 12 Months (n=1) | 100.0
  At 24 Months (n=3) | 66.7
  At 36 Months (n=2) | 100.0
  At 48 Months (n=1) | 100.0
  At 60 Months (n=1) | 100.0

33. Secondary Outcome: Percentage of Participants With Plasma HIV-1 RNA Levels Less Than 400 Copies/Milliliter [mL]) by Duration in Treatment-Experienced Participants
Description: as for outcome 32
Time Frame: Months 0, 3, 6, 9, 12, 24, 36, 48, and 60 after first dosing of Lopinavir/Ritonavir
Population: as for outcome 32
Measure: Number; unit: percentage of participants
Arm/Group | Lopinavir/Ritonavir
Number analyzed (Participants) | 4
percentage of participants
  At 0 Months (n=4) | 100.0
  At 3 Months (n=1) | 100.0
  At 6 Months (n=1) | 100.0
  At 9 Months (n=2) | 100.0
  At 12 Months (n=2) | 100.0
  At 24 Months (n=0) | NA — No data available for assessment.
  At 36 Months (n=0) | NA — No data available for assessment.
  At 48 Months (n=0) | NA — No data available for assessment.
  At 60 Months (n=0) | NA — No data available for assessment.

ADVERSE EVENTS:
Time Frame: Up to 60 Months
Arm/Group | Lopinavir/Ritonavir
Serious Adverse Events (participants affected / at risk) | 20/220
Other Adverse Events (participants affected / at risk) | 99/220
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Lopinavir/Ritonavir (N=220)
AMOEBIASIS (Infections and infestations) | 1
CHRONIC HEPATITIS C (Infections and infestations) | 1
LYMPH NODE TUBERCULOSIS (Infections and infestations) | 1
PULMONARY TUBERCULOSIS (Infections and infestations) | 1
MYCOBACTERIUM AVIUM COMPLEX INFECTION (Infections and infestations) | 1
ENTERITIS INFECTIOUS (Infections and infestations) | 1
HEPATITIS VIRUS-ASSOCIATED NEPHROPATHY (Infections and infestations) | 1
HERPES ZOSTER MENINGITIS (Infections and infestations) | 1
ANAL CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
HEPATIC CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
IMMUNE RECONSTITUTION INFLAMMATORY SYNDROME (Immune system disorders) | 1
CATARACT (Eye disorders) | 1
CARDIAC FAILURE (Cardiac disorders) | 1
PNEUMOTHORAX (Respiratory, thoracic and mediastinal disorders) | 1
INGUINAL HERNIA (Gastrointestinal disorders) | 1
LARGE INTESTINE POLYP (Gastrointestinal disorders) | 1
BILIARY COLIC (Hepatobiliary disorders) | 1
OSTEONECROSIS (Musculoskeletal and connective tissue disorders) | 2
NEPHROLITHIASIS (Renal and urinary disorders) | 1
THREATENED LABOUR (Pregnancy, puerperium and perinatal conditions) | 1
ABORTION INDUCED (Surgical and medical procedures) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Lopinavir/Ritonavir (N=220)
SYPHILIS (Infections and infestations) | 2
SKIN PAPILLOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
ANAEMIA (Blood and lymphatic system disorders) | 2
BASEDOW'S DISEASE (Endocrine disorders) | 1
HYPERTHYROIDISM (Endocrine disorders) | 1
DIABETES MELLITUS (Metabolism and nutrition disorders) | 2
HYPERCHOLESTEROLAEMIA (Metabolism and nutrition disorders) | 3
HYPERTRIGLYCERIDAEMIA (Metabolism and nutrition disorders) | 22
HYPERURICAEMIA (Metabolism and nutrition disorders) | 3
HYPOGLYCAEMIA (Metabolism and nutrition disorders) | 1
DYSLIPIDAEMIA (Metabolism and nutrition disorders) | 2
HYPERPHOSPHATASAEMIA (Metabolism and nutrition disorders) | 4
LIPID METABOLISM DISORDER (Metabolism and nutrition disorders) | 1
HYPERLIPIDAEMIA (Metabolism and nutrition disorders) | 15
HYPO HDL CHOLESTEROLAEMIA (Metabolism and nutrition disorders) | 1
DEPRESSION (Psychiatric disorders) | 5
INSOMNIA (Psychiatric disorders) | 5
CERVICOBRACHIAL SYNDROME (Nervous system disorders) | 1
HEADACHE (Nervous system disorders) | 2
HYPOAESTHESIA (Nervous system disorders) | 1
SCIATICA (Nervous system disorders) | 1
CONJUNCTIVITIS ALLERGIC (Eye disorders) | 1
CORNEAL EROSION (Eye disorders) | 1
CHORIORETINOPATHY (Eye disorders) | 1
DEAFNESS (Ear and labyrinth disorders) | 1
TINNITUS (Ear and labyrinth disorders) | 1
CONGESTIVE CARDIOMYOPATHY (Cardiac disorders) | 1
HYPERTENSION (Vascular disorders) | 2
ASTHMA (Respiratory, thoracic and mediastinal disorders) | 2
RHINITIS ALLERGIC (Respiratory, thoracic and mediastinal disorders) | 1
ABDOMINAL PAIN (Gastrointestinal disorders) | 1
CONSTIPATION (Gastrointestinal disorders) | 1
DIARRHOEA (Gastrointestinal disorders) | 9
GASTRITIS (Gastrointestinal disorders) | 1
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 2
NAUSEA (Gastrointestinal disorders) | 1
HEPATIC FUNCTION ABNORMAL (Hepatobiliary disorders) | 4
HYPERBILIRUBINAEMIA (Hepatobiliary disorders) | 1
LIVER DISORDER (Hepatobiliary disorders) | 6
DRUG-INDUCED LIVER INJURY (Hepatobiliary disorders) | 1
ACNE (Skin and subcutaneous tissue disorders) | 1
DERMATITIS (Skin and subcutaneous tissue disorders) | 1
PRURITUS (Skin and subcutaneous tissue disorders) | 1
RASH (Skin and subcutaneous tissue disorders) | 1
URTICARIA (Skin and subcutaneous tissue disorders) | 1
LIPODYSTROPHY ACQUIRED (Skin and subcutaneous tissue disorders) | 1
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 1
POLYARTHRITIS (Musculoskeletal and connective tissue disorders) | 1
OSTEOPENIA (Musculoskeletal and connective tissue disorders) | 1
CALCULUS URETERIC (Renal and urinary disorders) | 1
CALCULUS URINARY (Renal and urinary disorders) | 1
NEPHROLITHIASIS (Renal and urinary disorders) | 1
RENAL DISORDER (Renal and urinary disorders) | 1
RENAL IMPAIRMENT (Renal and urinary disorders) | 5
GYNAECOMASTIA (Reproductive system and breast disorders) | 1
PYREXIA (General disorders) | 1
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 1
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 1
BETA 2 MICROGLOBULIN URINE INCREASED (Investigations) | 17
BLOOD BILIRUBIN INCREASED (Investigations) | 1
BLOOD CREATINE PHOSPHOKINASE INCREASED (Investigations) | 1
BLOOD CREATININE INCREASED (Investigations) | 2
BLOOD TRIGLYCERIDES INCREASED (Investigations) | 13
BLOOD URIC ACID INCREASED (Investigations) | 3
C-REACTIVE PROTEIN INCREASED (Investigations) | 1
GAMMA-GLUTAMYLTRANSFERASE INCREASED (Investigations) | 13
GLUCOSE URINE PRESENT (Investigations) | 1
HAEMOGLOBIN DECREASED (Investigations) | 1
LIPIDS ABNORMAL (Investigations) | 2
LOW DENSITY LIPOPROTEIN INCREASED (Investigations) | 1
RED BLOOD CELL COUNT DECREASED (Investigations) | 1
WHITE BLOOD CELL COUNT INCREASED (Investigations) | 1
PROTEIN URINE PRESENT (Investigations) | 2
TRANSAMINASES INCREASED (Investigations) | 1
BLOOD ALKALINE PHOSPHATASE INCREASED (Investigations) | 8
HEPATIC ENZYME INCREASED (Investigations) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.